CLINICAL TRIAL: NCT05809908
Title: A Phase 3, 26-Week, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of Daily Administration of Tricaprilin as AC-OLE-01-VA in Participants With Mild to Moderate Alzheimer's Disease Dementia
Brief Title: Tricaprilin Phase 3 ALTER-AD (Alternative-Alzheimer Disease) Study
Acronym: ALTER-AD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-22-027
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tricaprylin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tricaprilin (Active Comparator): Tricaprilin formulation twice daily for 26 weeks, liquid for oral administration
  Interventions: Drug: Tricaprilin
- Placebo (Placebo Comparator): Placebo formulation, twice daily for 26 weeks, liquid for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tricaprilin — Each dose of IMP will be administered orally 30 minutes after completing a full meal.
  There is 1 g of tricaprilin per 2 ml of AC-OLE-01-VA.
  Participants will titrate from 5 g twice a day to 20 g twice a day, up to 40 g total daily dose of tricaprilin; 80 ml total daily dose of AC-OLE-01-VA, over the course of 2-4 weeks.
  Arms: Tricaprilin
Drug: Placebo — Each dose of IMP will be administered orally 30 minutes after completing a full meal.
  Participants will titrate from 5 g twice a day to 20 g twice a day, up to 40 g total daily dose of placebo; 80 ml total daily dose of placebo, over the course of 2-4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of tricaprilin (20 g twice a day) on cognition, global function, activities of daily living, resource utilisation, safety, and tolerability, in participants with mild to moderate AD dementia.

This is a randomised, double-blind, placebo-controlled, parallel-group, multi-centre design in up to 535 participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Mini Mental State Exam (MMSE) score between 14 to 24
* Meets diagnostic clinical criteria of probable Alzheimer's disease dementia according to the NIA-AA criteria
* Magnetic resonance imaging (MRI) scan less than 12 months before Baseline compatible with a diagnosis of probable AD
* Plasma biomarker result supporting a diagnosis of AD before Baseline (Aβ42/40 and/or pTau217)
* Confirmed APOE4 genotype result prior to Baseline
* Participants taking the following cholinesterase inhibitors: donepezil, galantamine, or rivastigmine; and/or sodium oligomannate (GV-971), and/or memantine, and/or GLP-1 antagonist and/or other agents which may impact cognition are eligible for enrolment: a) If the participant has been taking such medication(s)/products for 3 months or more at Screening Visit 1; b) If the current dosage regimen is within the approved dose range; c) The daily dose has remained unchanged for at least 6 weeks prior to screening; d) If the dose is not expected to change during study participation

Key Exclusion Criteria:

* Has any medical/neurological/psychiatric condition, other than AD, that could explain the participant's dementia or cognitive impairment, such as but not limited to e.g., structural abnormality, traumatic brain injury, stroke, epilepsy, Parkinson's disease, alcohol-related dementia, current major depressive episode
* The following GI conditions are exclusionary: a) Inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), GI bleed (upper or lower), or peptic ulcer disease; any of these conditions are exclusionary, if active in the past 5 years. Participants with remote quiescent disease, at the Investigators discretion , are not excluded; b) Participants with current or a history of (within the last 5 years) any of the following conditions are excluded: clinically significant reflux disease (e.g., Barrett's oesophagus, stricture, ulcer, haemorrhage), or severe gastroesophageal reflux disease that, in the opinion of the Investigator, is not well-controlled by medication; c) Irritable bowel syndrome, diverticular disease (e.g., diverticulosis, or diverticulitis), or chronic gastritis; any of these conditions are exclusionary if there has been an acute event within 1 year prior to Screening; d) History of gastric food intolerance, whether it be allergy or chronic oversensitivity, or a history of stomach upset reaction to a variety of foods
* Current or previous treatment with any anti-amyloid or anti-Tau antibodies such as lecanemab and donanemab within 6 months prior to the day of screening

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) total score | 26 weeks
  The ADAS-Cog is a cognitive scale that assesses memory, language, orientation, and praxis with a total score range of 0 (no impairment) to 70 (severe impairment).
Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | 26 weeks
  The ADCS-CGIC is a clinician-rated scale of cognition, function, and behavior. Scores range from 1 (marked improvement) to 7 (marked worsening).

SECONDARY OUTCOMES:
Change From Baseline in a composite score of Category Fluency Test (CFT), Controlled Oral Word Association Test (COWAT), and ADAS-Cog subtests Word Recall, Word Recognition and Orientation | 26 weeks
  The CFT is a cognitive test assessing a participant's semantic fluency, a measure of executive function. Participants are given 60 seconds to name as many examples of a category, with 1 point for each correct, unique response given.
  The COWAT is a cognitive test assessing a participant's phonemic fluency, a measure of executive function. Participants are given 60 seconds (per word) to say as many words as possible beginning e.g., with the letters F, A and S (in English, equivalents will be used for other languages), with 1 point for each original and correct word.
  The ADAS-Cog is a cognitive scale that assesses memory, language, orientation, and praxis with a total score range of 0 (no impairment) to 70 (severe impairment).
Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score | 26 weeks
  The ADCS-ADL is a 23-item semi-structured interview with a caregiver and assesses 6 basic activities of daily living and 7 instrumental activities of daily living with a total score of 0 to 78. Lower scores indicate greater severity.

OTHER OUTCOMES:
Exploratory Biomarker Analysis | 26 weeks
  * Change in glial fibrillary acidic protein (GFAP) and neurofilament light chain protein (NfL) biomarker levels from Baseline to Week 26.
  * Change in plasma Aβ biomarker levels from Baseline to Week 26.
  * Change in phosphorylated tau biomarker levels from Baseline to Week 26.
  * Change in validated metabolomics biomarker levels from Baseline to Week 26.